CLINICAL TRIAL: NCT04269863
Title: Personalizing Antiplatelet Therapy in Peripheral Arterial Disease Patients
Brief Title: Personalizing Aspirin Therapy in Peripheral Arterial Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Mohammad, Vascular Surgeon, Unity Health Toronto
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-241
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Aspirin
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: 150 patients randomized into two groups of 75 patients each, one control group receiving 81mg ASA and treatment group receiving a personalized dose of unto 325mg (within the recommended dosage limits)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): This group of 75 patients is the control group that will be receiving the standard lowest dosage of 81mg aspirin.
  Interventions: Drug: Aspirin
- Treatment Group (Experimental): This group of 75 participants is the treatment group that will be receiving personalized aspirin dosage between 81mg-325mg (within standard clinical recommendations), which will be determined based on platelet analysis via PFA-200.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — control - 81mg. treatment - 81-325mg.

SUMMARY:
Antiplatelet therapies are important to decrease the morbidity and mortality associated with Peripheral Arterial Disease (PAD) through the prevention of thrombus formation. Aspirin (ASA) is a readily available and affordable antiplatelet medication that can help reduce adverse cardiovascular events by up to 25%. However, 25-60% of PAD patients are "ASA insensitive" having a lower than normal ability to inhibit platelet aggregation after standard aspirin dosing. In a previous study conducted by our lab, we were able to demonstrate a methodology for personalizing antiplatelet therapy using two platelet function tests, Platelet Function Analyzer-100 (PFA 100) and Light Transmission Aggregometry (LTA). To investigate this methodology further, we would like to conduct a pilot study on two cohorts of patients, one population continuing with their current medications (81mg ASA), and a second group who will get personalized antiplatelet therapy using our methodology (81-325mg ASA). In this study, 150 PAD patients taking 81mg Aspirin therapy presenting for clinical follow-up, or in-patient intervention, in vascular clinics or the emergency room, will be recruited to our study. 75 patients will be randomly assigned undergo platelet analysis using PFA-200 and LTA, and will have their antiplatelet therapy personalized. Patients will then be followed up in order to see if the patients with personalized therapy have better platelet inhibition. This study will allow us to help personalize antiplatelet therapy in PAD patients, allowing for better patient outcomes and decreased adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported intake of either 81 mg of aspirin per day for 3 or more days
* Diagnosed with peripheral arterial disease

Exclusion Criteria:

* Alcohol ingestion 24 hours prior to blood draw
* Patients receiving glycoprotein (GP) IIb/IIIa antagonists
* Ingestion of a non steroidal anti-inflammatory drug 3 days prior to blood draw
* History of bleeding disorders
* Gastrointestinal bleeding
* Hemorrhagic stroke
* Allergy to aspirin or ticagrelor
* Pregnancy, thrombocytopenia anmia or leukopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
PAD disease progression | 1 year
  Using lower limb arterial imaging (doppler ultra sound), and ankle brachial index, patients will be categorized based on Ruthorford Classification of chronic limb ischemia. Progression of PAD will be considered decrease in ABI, and progression to more sever forms according to the Rutherford classification.
development of Critical limb ischemia | 1 year
  Critical limb ischemia will considered as those patients who have progressed from claudication to night paint, rest pain, and/or tissue loss.

IPD SHARING:
Plan to Share IPD: No